CLINICAL TRIAL: NCT04516239
Title: Prospective Double-blind Randomized Clinical Trial Comparing Gait Analysis and Clinical Function After Metal on Metal Total Hip Arthroplasty With Large Diameter Femoral Head and Metal on Metal Total Hip Resurfacing.
Brief Title: Comparison of Metal on Metal Total Hip Arthroplasty and Metal on Metal Total Hip Resurfacing.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Pascal-André Vendittoli, Orthopedist, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04132
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Arthroplasty; Replacement; Hip
Keywords: Metal-Metal; Large Diameter Head Total Hip Arthroplasty; Hip Resurfacing

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized clinical trial with two parallel treatment groups. At the preoperative teaching session, the study objectives and the risks and benefits of surgery will be explained to the patient by the research assistant or the surgeon in order to obtain consent. A randomization table will be generated by the SPSS 10 software and sealed numerated envelopes will be assigned to each patient entering the study. A research assistant will coordinate the study and data collection.
Who Masked: Participant
Masking Description: The patient will be informed of the randomization group, 6 months after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDH THA (Active Comparator): large diameter head total hip arthroplasty
  Interventions: Device: THA
- HR (Active Comparator): metal-on-metalhip resurfacing
  Interventions: Device: HR

INTERVENTIONS:
Device: THA — Three surgeons performed the surgeries through a posterior surgical approach in both groups. The fascia lata was opened and the gluteus maximus was split in line with its muscle fibers. The short external rotators were released from the greater trochanter. A posterior capsulotomy was performed and the hip dislocated. For the THA, the standard techniques proposed by the manufacturer for insertion of the stem were followed. Neck sleeve adapters and three different prosthetic neck-shaft angles (125, 135, and 145) were available to adjust leg length and femoral offset with the large-diameter head THA system.
  Arms: LDH THA
Device: HR — Three surgeons performed the surgeries through a posterior surgical approach in both groups. The fascia lata was opened and the gluteus maximus was split in line with its muscle fibers. The short external rotators were released from the greater trochanter. A posterior capsulotomy was performed and the hip dislocated. In the HR group, the capsulotomy was completed circumferentially, and the gluteus tendinous insertion on the femur was released in all men, but only when needed in women, to improve femur mobilization.
  Arms: HR

SUMMARY:
The goal of this double-blind prospective randomized study is to compare subjective outcome measures and gait parameters between conventional THA using large diameter femoral heads and total hip resurfacing

DETAILED DESCRIPTION:
In the early 1960's Sir John Charnley revolutionized total hip arthroplasty (THA) with the introduction of polyethylene as a bearing surface. This innovation allowed THA to become a very successful procedure to treat degeneration of the hip joint, with excellent long term clinical outcome and patient satisfaction.

However, this technique requires sacrifice of the whole femoral head and part of the neck. This bone will not be available for future revision surgery, which seems inevitable in the younger patient. THA does not always allow precise reconstitution of normal hip biomechanics. The femoral canal is also violated, fat and cement embolism can occur and thrombogenic material is released in the bloodstream. Postoperatively the femoral stem can cause thigh pain, proximal stress shielding, and periprosthetic fracture may occur . Finally the use of a 28 millimeter non anatomic femoral head during conventional THA increases the risk of hip impingement and dislocation while limiting hip range of motion.

There is renewed interest in the concept of hip resurfacing and the use of large diameter femoral heads in total hip arthroplasty, since both these options recreate more optimal hip biomechanics. Total hip resurfacing is less invasive than conventional THA using a femoral stem and allows restoration of normal hip anatomy. Additionally, compared to conventional THA, hip resurfacing has the following advantages: preservation of the femoral head and neck, better hip stability, improved hip biomechanics (leg length, offset) and possibly better proprioception. Since the femoral canal is not violated, there is less risk of residual thigh pain, and patients probably have the sensation of a more normal feeling joint.

As for conventional THA with large diameter femoral heads, the use of a near anatomic head size (compared to the small 28mm diameter head use with conventional THA) restores normal stability, helps reduce the incidence of impingement and increases range of motion to a greater extent than hip resurfacing, and might improve proprioception as well. The investigators believe these advantages will have a positive influence on clinical function and gait pattern compared to conventional THA.

Gait analysis has demonstrated that gait pattern is modified after THA and patients do not recover normal gait. Kinematics analysis further showed that abnormal gait pattern is not only observed in the operated hip but also in other articulations, including the contra lateral limb. Walking kinetics are affected to some extent, especially the force generated by the lower limb and synchronization of muscle activity. Finally a subjective feeling of an abnormal hip function may still persists after THA.

The goal of this double-blind prospective randomized study is to compare subjective outcome measures and gait parameters between conventional THA using large diameter femoral heads and total hip resurfacing

ELIGIBILITY:
Inclusion Criteria:

1. Patient with degenerative disease of the hip in need for total hip or total hip resurfacing arthroplasty
2. Patient who understands the study protocol and willing to comply with the planned clinical follow-up
3. Patient can give informed consent

Exclusion Criteria:

1. Age older than 65 years old or younger than 18 years old
2. Charnley class B (both hip diseased) or C (polyarticular disease) patients
3. Spinal or lower limb disease other than the degenerated hip that could influence gait and walking performance
4. Neuromuscular disorder
5. Known or suspected metal allergy
6. Pregnancy
7. Renal insufficiency
8. Known or suspected osteopenia or osteoporosis of the hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Implant revisions | Preoperative to 15 years
  Implant revisions rate will be compared between groups.
Reasons of revisions | Preoperative to 15 years
  Reasons of revisions will be categorized and compared between groups.
Adverse events | Preoperative to 15 years
  Adverse events will be categorized and compared between groups.

SECONDARY OUTCOMES:
Patient reported outcome measures (PROMs) : Womac | Preoperative to 15 years
  Womac score will be compared between groupsScore and Patient's Joint Perception.
Patient reported outcome measures (PROMs) : UCLA activity | Preoperative to 15 years
  The UCLA activity score will be compared between groups.
Patient reported outcome measures (PROMs) : Forgotten Joint | Preoperative to 15 years
  Forgotten Joint score will be compared between groups.
Whole blood chromium metal ions levels | Preoperative to 15 years
  Whole blood chromium metal ion measurements will be compared between groups for participants without other bodily metallic implants or revised implants.
Whole blood cobalt metal ions levels | Preoperative to 15 years
  Whole blood cobalt metal ion measurements will be compared between groups for participants without other bodily metallic implants or revised implants.
Radiological evaluation of femoral stem loosening | Preoperative to 15 years
  Signs of definite femoral stem loosening included continuous lucent lines > 2 mm, stem fracture, subsidence > 5 mm, or a change in component angulation >5° will be compared between groups.
Radiological evaluation of acetabular loosening | Preoperative to 15 years
  Signs of definite acetabular loosening presented as continuous radiolucency > 2 mm, component migration > 3 mm or angulation change >5° will be compared between groups.
Radiological evaluation of heterotopic ossification | Preoperative to 15 years
  Signs of heterotopic ossification grade, estimated according to the Brooker classification, will be compared between groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kostretzis L, Lavigne M, Kiss MO, Shahin M, Barry J, Vendittoli PA. Despite higher revision rate, MoM large-head THA offers better clinical scores than HR: 14-year results from a randomized controlled trial involving 48 patients. BMC Musculoskelet Disord. 2021 Apr 30;22(1):400. doi: 10.1186/s12891-021-04286-6. PMID 33941155
- See also: The John Charnley Award: The functional outcome of hip resurfacing and large-head THA is the same: a randomized, double-blind study — https://pubmed.ncbi.nlm.nih.gov/19543863/